CLINICAL TRIAL: NCT02043899
Title: A Cancer Research UK Phase I/II Study to Compare [124I]Meta-Iodobenzylguanidine (mIBG) Positron Emission Tomography/Computerised Tomography (PET/CT) to [123I]mIBG Imaging in Patients With Metastatic Neuroblastoma
Brief Title: A Phase I/II Study of [124I]mIBG PET/CT in Neuroblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRUKD/12/002; 2012-002029-31 (EudraCT Number)
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Results first posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-05

CONDITIONS: Metastatic Neuroblastoma
Keywords: Neuroblastoma; Positron emission tomography; 124-iodine; Meta-Iodobenzylguanidine
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Trial (Experimental): This was a single arm trial, all patients were to undergo the same assessments and interventions.
  Interventions: Drug: [124I]meta-Iodobenzylguanidine

INTERVENTIONS:
Drug: [124I]meta-Iodobenzylguanidine — Single intravenous administration of [124I]mIBG Solution for Injection on Day 1 with a maximum radioactive dose of 1.42 MBq/kg (±10%) and a maximum injected dose of 50 MBq [124I]mIBG equating to a maximum chemical dose of 10 micrograms of stable mIBG. The activity to paediatric patients will be scaled by weight based upon the EANM paediatric dose card (Lassmann et al., 2007). This will result in an activity between 10 MBq and 50 MBq depending on the patient's weight.

SUMMARY:
This study aims to show that 3-dimensional PET/CT imaging with a new novel PET tracer (called [124I]mIBG) can detect as many or more sites of neuroblastoma (a type of childhood cancer) compared to the recommended 1-dimensional routine scans (called [123I]mIBG planar scintigraphy).

DETAILED DESCRIPTION:
Neuroblastoma is the most common tumour of childhood after brain tumours. Approximately half of cases are high risk and despite extensive treatments outcome is very poor. More than 60% of high risk patients suffer relapse or further spread of their disease and long-term survival is below 10%. Existing imaging techniques are not sensitive enough to accurately assess the level of risk which is critical in determining the best choice of treatment. This study will compare a new type of imaging against the existing imaging techniques. The new scans use a new tracer called [124I]mIBG which is taken up by the cancer tissue much more than by normal tissues. This tracer can be used with a 3D imaging technique called PET/CT to pinpoint where the disease has spread and quantify the amount of disease. Patients will be those scheduled to have an [123I]mIBG scan for routine care during a planned break in treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven Stage 4 neuroblastoma as defined by the International Neuroblastoma Staging System (INSS).
2. Aged ≥ 1 year at the time that written informed consent is given.
3. Planned to undergo conventional [123I]mIBG planar scintigraphy for routine clinical care of neuroblastoma.
4. Life expectancy of at least 12 weeks.
5. World Health Organisation (WHO) performance status of 0, 1 or 2 for patients aged > 12 years old or Lansky play scale score of ≥ 50% for patients aged ≤ 12 years old.
6. Written (signed and dated) informed consent from patient ≥ 16 years old and/or parent or legal guardian for patients <16 years old and the patient be capable of co-operating with scanning requirements. (N.B. Written or verbal assent as appropriate should be sought from all patients who are under 16 years old).

Exclusion Criteria:

1. Treatment with any medications contra-indicated with mIBG scanning as listed in Appendix 4 of the trial protocol. For example, decongestants containing pseudoephedrine, phenylpropalomine and phenylephrine, sympathomimetics, cocaine, antihypertensives, tricyclic antidepressants. These drugs should be stopped before administration as indicated in this list (usually for four biological half-lives to allow almost complete wash-out but refer to list).
2. Stage 4S neuroblastoma as defined by the INSS.
3. Any anti-cancer treatment planned between the routine [123I]mIBG imaging and the [124I]mIBG PET/CT scan on Day 2. Anti-cancer treatments can be started only after the Off-Study assessment on Day 3 to Day 7, see schedule of assessments in Section 7. N.B. Patients should not be enrolled in the study if their participation will delay their subsequent treatment for neuroblastoma.
4. Female patients who are pregnant or lactating.
5. At high medical risk because of non-malignant systemic disease including active uncontrolled infection.
6. Known to be serologically positive for Hepatitis B, Hepatitis C or Human Immunodeficiency Virus (HIV).
7. Patients with known hypersensitivity to mIBG.
8. Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical study.

Clinical Criteria for [124I]mIBG imaging

1. One or more disease foci observed on conventional [123I]mIBG planar scintigraphy. Disease foci will initially be identified by a Nuclear Medicine physician at the investigational site.
2. ≥ 3kg at the time of the [124I]mIBG imaging to agree with the paediatric EANM guidelines.
3. Haematological and biochemical indices within the ranges below:

   For patients ≤16 years old, haematological and biochemical indices within the following ranges: Haemoglobin ≥ 7.0 g/dl (N.B transfusions will be allowed); Absolute neutrophil count ≥ 0.2 x 10^9/L (N.B. G-CSF support will be allowed); Platelet count ≥ 10 x 10^9/L (N.B. transfusions will be allowed); Serum bilirubin ≤ 2.5 x upper limit of normal (ULN); Alanine amino-transferase (ALT), aspartate amino-transferase (AST), and/ or alkaline phosphatase (ALP) ≤ 5 x ULN; and Calculated creatinine clearance using revised Schwartz formula ≥ 60 mL/min/1.73m^2.

   For patients >16 years old, haematological and biochemical indices within the following ranges: Haemoglobin ≥ 8.0 g/dl (N.B transfusions will be allowed); Absolute neutrophil count ≥ 0.5 x 10^9/L (N.B. G-CSF support will be allowed); Platelet count ≥ 50 x 10^9/L (N.B. transfusions will be allowed); Serum bilirubin ≤ 2.5 x upper limit of normal (ULN); Alanine amino-transferase (ALT), aspartate amino-transferase (AST), and/ or alkaline phosphatase (ALP) ≤ 5 x ULN; and Estimated Glomerular Filtration Rate (eGFR) ≥ 60 mL/min/1.73m^2.
4. Menarchal female patients must have a negative serum or urine pregnancy test before administration of [124I]mIBG Solution for Injection on Day 1 and agree to use two highly effective forms of contraception (oral, injected or implanted hormonal contraception and condom, have an intra-uterine device and condom, diaphragm with spermicidal gel and condom) to be effective from Day 1 and for 7 days afterwards.
5. Male patients with partners of child-bearing potential must agree to take measures not to father children by using one form of highly effective contraception [condom plus spermicide] from Day 1 and for 7 days afterwards. Male patients with pregnant or lactating partners must agree to use barrier method contraception (e.g. condom plus spermicidal gel) to prevent exposure to the foetus or neonate.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Chua, Dr, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - University College London Hospital, London
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial participants were enrolled at two trial sites between 11 February 2014 and 10 September 2019.
Period: Overall Study
Arm/Group | Single Arm Trial
Started | 36
Underwent Routine [123I]mIBG Planar and SPECT/CT Imaging | 32
Underwent [124I]mIBG PET/CT Imaging | 9
Completed | 9
Not Completed | 27
Not completed — Adverse Event | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2
Not completed — Failure to meet the clinical criteria for [124I]mIBG imaging | 5
Not completed — Technical manufacturing issue or logistical difficulties of [123I]mIBG or [124I]mIBG supply | 12
Not completed — Temporary halt due to out of specification radioactivity | 2
Not completed — Clinical progression necessitating urgent treatment | 1
Not completed — Treatment delayed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 36

OUTCOME MEASURES:

1. Primary Outcome: Comparison of the Number of Lesions Detected as Positive by [123I]mIBG Planar Scintigraphy Which Are Also Considered Positive With [124I]mIBG PET/CT.
Description: Analysis of [124I]mIBG PET/CT and [123I]mIBG planar scintigraphy was performed retrospectively by four specialist observers. The analysis was performed and observers were blinded to each others scores. The observers subsequently reviewed the lesions identified and, where there was a difference in their separate scores, they returned to the images in order to reach an agreed consensus score. The number of lesions identified as positive by this consensus scoring (all lesions with a SIOPEN score of 4 or 5) were used to meet the primary objective.
Time Frame: [124I]mIBG PET/CT imaging on Day 1, three to 21 days after routine [123I]mIBG imaging and before the start of any new anti-cancer therapy. A minimum interval of 72 hours was required between injection of [123I]mIBG tracer and the [124I]mIBG PET/CT scan.
Population: All patients who received both [123I]mIBG and [124I]mIBG
Measure: Number; unit: Lesions
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 9
Lesions
  Number of positive lesions observed using [124I]mIBG PET/CT | 714
  Number of positive lesions observed using [123I]mIBG planar scintigraphy | 405
Statistical Analysis 1: Comparison: Single Arm Trial; Test type: Other — 1. Exact one-sided binomial test of the null hypothesis (p≤90%) using α=0.05 on [124I]mIBG PET/CT SIOPEN consensus scores. If this was accepted and the alternative hypothesis rejected, then trial stopped early for futility. 2. If the null hypothesis was rejected, then a one-sided binomial test of the null hypothesis (p≥97%) was performed (α=0.025). If this was accepted and the alternative hypothesis rejected then the trial stopped early for efficacy; p < 0.001, Exact one-sided binomial test — Overall design has 82% power and an α of 0.03. Total minimum sample size of 100 lesions was calculated based on a single stage A'hern design with p0 = 0.90 and p1 = 0.97. The overall power and α was calculated based on exact binomial probabilities; For the primary endpoint, a sensitivity analysis was also performed on patients with <20 positive lesions on [124I]mIBG PET/CT to test if few patients with large numbers of positive lesions were affecting the results. The results of the sensitivity analysis were consistent with those of the overall analysis. Secondary efficacy analysis, separate exact one-sided binomial test of the null hypothesis (p≥97%), performed (α=0.025) performed for skeletal and soft tissue lesions

2. Secondary Outcome: Comparison of the Number of Lesions Detected as Positive by [123I]mIBG SPECT Which Are Also Considered Positive With [124I]mIBG PET/CT.
Description: Analysis of [124I]mIBG PET/CT and [123I]mIBG SPECT/CT was performed retrospectively by four specialist observers. The analysis was performed and observers were blinded to each others scores. The observers subsequently reviewed the lesions identified and, where there was a difference in their separate scores, they returned to the images in order to reach an agreed consensus score. The number of lesions identified as positive by this consensus scoring (all lesions with a SIOPEN score of 4 or 5) were used to meet the primary objective.
Time Frame: as for outcome 1
Population: All patients who received both [123I]mIBG and [124I]mIBG
Measure: Number; unit: Lesions
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 9
Lesions
  Number of positive skeletal lesions observed using [124I]mIBG PET/CT | 421
  Number of positive skeletal lesions observed using [123I]mIBG SPECT/CT | 249
  Number of positive soft tissue lesions observed using [124I]mIBG PET/CT | 132
  Number of positive soft tissue lesions observed using [123I]mIBG SPECT/CT | 64

3. Secondary Outcome: Determining the Causality of Each Adverse Event to [124I]mIBG and Grading Severity According to National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) Version 4.02.
Description: Documenting Adverse Events (AEs), Serious Adverse Events (SAEs), Dose Limiting Toxicities (DLTs) (Graded According to NCI-CTCAE Version 4.02) and Laboratory Parameters and Determining Their Causality in Relation to [123I]mIBG and [124I]mIBG.
Time Frame: Safety data was collected from the date of written informed consent and continued for seven days after administration of [124I]mIBG.
Measure: Number; unit: Events
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 32
Events
  All AEs | 25
  Pretreatment AEs (occurring before [123I]mIBG administration) | 16
  Treatment Emergent AEs (occurring following [123I]mIBG administration) | 9
  SAEs | 3
  [123I]mIBG Related AEs | 0
  [124I]mIBG Related AEs | 0

ADVERSE EVENTS:
Time Frame: Safety data was collected from the date of written informed consent and continued for seven days after administration of [124I]mIBG.
Arm/Group | Single Arm Trial
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 2/32
Other Adverse Events (participants affected / at risk) | 10/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Trial (N=32)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) — Verbatim term new central line Insertion (surgical procedure) due to central line being accidentally removed.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Trial (N=32)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Ear Pain (Ear and labyrinth disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Oral pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Fever (General disorders) | 2 (2)
Mucosal infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1) — Verbatim term: sore vulval region
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
An exact one-sided binomial test of the null hypothesis: p ≤90% was performed using α=0.05 on the [124I]mIBG PET/CT imaging assessments with SIOPEN consensus scores.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT02043899/Prot_SAP_000.pdf